CLINICAL TRIAL: NCT05846074
Title: Pilot Study for the Experimental Validation of the Intrinsic Diagnostic Performance Among the First Dod Team for the Canine Olfactory Detection of COVID-19 on Sweat Samples From Persons Tested by PCR SARS-CoV-2.
Brief Title: Diagnostic Performance of Dogs for the Olfactory Detection of COVID-19
Acronym: CYNOCOV
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/05
Record Dates: First submitted 2023-05-04; First posted 2023-05-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: COVID-19; dog; canine; olfactory; diagnostic
MeSH Terms: conditions — COVID-19; Anosmia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of sweat samples and face mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sweat samples and used face mask will be collected — Collection of sweat samples and used face mask will take approximately 15 minutes before or after collection for the SARS-Cov PCR test

SUMMARY:
Considering the favorable preliminary data of few european diagnostic studies on dog detection, we develop in 2021 a pilot study in response to the plan of CHU Bordeaux and Nouvelle Aquitaine French region for an expanded, reliable and alternative rapid dog olfactory detection of COVID during pandemic period.

Our hypothesis is that validated olfactory detection on sweat or face mask collection by dogs would increase the acceptability and propensity to be tested in different population groups, given the non-invasive nature of sweat and face mask; compared to the unpleasant aspect of nasal swabs for PCR or rapid antigenic tests.

To reach this objective, we recruited a dog team to be trained and assessed (all-volunteers masters and dogs) and we will recruit participants with positive and negative PCR test. The diagnostic performance of canine olfactory detection of COVID-19 on sweat and face collection will be compared to the nasal SARS-Cov-2 PCR test of the participants.

DETAILED DESCRIPTION:
The design of the study is an open,interventional risk-free, multi-centre diagnostic validation pilot sudy The main objective is the experimental assessment of the intrinsic diagnostic performance (sensitivity, specificity) among the first dog team in Nouvelle Aquitaine French region for the canine olfactory detection of COVID-19 on sweat samples from persons tested by PCR SARS-CoV-2.

The secondary objectives are :

* the experimental assessment of the intrinsic diagnostic performance (sensitivity, specificity) according to different factors: symptomatic or not, comorbidity, gender, hormonal cycle of women, medication taking, anti-COVID-19 vaccination, canine characteristics and canine detection procedures.
* Proof of concept of canine olfactory detection performance with a used face mask.
* Determine the biochemical composition of the volatile organic compound(s) (VOCs) associated with COVID-19 and detected by the dogs team.
* the assessment of intrinsic and discriminating diagnostic performance (positive and negative predictive values) of dogs for the olfactory detection of COVID-19 on used sweat and/or face mask based on the symptomatology.

This study will be conducted in two phases:

- Phase 1: experimental assessment of the intrinsic diagnostic performance (sensitivity, specificity) among the first dogs team in Nouvelle Aquitaine French region for the canine olfactory detection of COVID-19 on sweat samples and face mask from persons tested by PCR SARS-CoV-2.

The experimental assessment of the phase 1 wil include two experimental subpopulation samples of people tested by PCR SARS-CoV-2: positive, symptomatic or non-symptomatic (Case subpopulation); and negative non-case-contact, symptomatic or non-symptomatic (Control subpopulation).

- Phase 2: Near-routine live assessment of intrinsic and discriminating diagnostic performance (positive and negative predictive values) of dogs for the olfactory detection of COVID-19 on sweat collection and/or used face mask of persons rountinely screened by PCR SARS-CoV-2. These persons will be recruited consecutively without discrimination of subpopulations.

ELIGIBILITY:
Inclusion Criteria:

* Criteria inclusion for "Case" participant Positive SARS-CoV-2 PCR test with significant viral load according to Ct <37 (high-speed extractor MGISP-960; used in CHU Bordeaux) or <34 (excluding high-speed extractor MGISP-960) Symptomatic person for a maximum of 7 days at the time of the sweat sample; or asymptomatic person with sweat sample within 72 hours of the PCR test.
* Criteria inclusion for witnessesControl participant Totally negative SARS-Cov-2 PCR test with sweat sampling within 72 hours Systematic screening (except in case of COVID-19 pre-contact ): air flight or surgical operation or unusual meeting or symptomatology or collective screening at the request of an organization Asymptomatic person (no unusual symptoms) for at least 1 month or unusual symptoms for at least of 48 hours and at mostof 5 days at the time of the PCR test

Exclusion Criteria:

-Common non-inclusion criteria: Age less than 6 years old History of COVID-19 confirmed by PCR test or rapid test or Scanner between Day 8 and Day 35 of the onset of symptoms -or of the test if asymptomatic) History of taste and / or smell disorder (s) that occurred between the Day 8 and Day 35 before pre-inclusion.

Confirmed or suspected long-haul symptoms of COVID-19 Patient subject to a judicial protection measure Person opposing the study (child or parent if minor) OR not understanding French

-Criteria for non-inclusion of witnessesControl participant : Contact case of COVID-19 for less than 35 days without having made PCR test between Day 5 and Day 8 of the contact Vaccination date against COVID of 7 days or less Professionals in human health or nursing homes or medical transport Woman in the middle of the menstrual cycle without pill or implant type contraception (ovulation) History of taste and / or smell disorders that occurred less than 7 days ago Hospitalization for more than 724 hours at the time of the sweat collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people screened by SARS-CoV2 PCR
Sampling Method: Non-Probability Sample
Enrollment: 1548 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Experimentally validate the intrinsic diagnostic performance of dogs for the olfactory detection of COVID-19 | day 1
  Combined measurement of a Sensitivity > 80% and a specificity > 60% of each dog and of all the dogs eligible for the week of evaluation of the canine olfactory detection of COVID-19; compared to the SARS-Cov-2 PCR test (gold standard)

SECONDARY OUTCOMES:
Experimentally validate the intrinsic performance | day 1
  Combined measurement of Sensitivity > 80% and Specificity > 60% of each dog and of all dogs eligible for the week of evaluation; in different subgroups of participants according to the presence of symptomatology, the presence of comorbidities, gender, hormonal cycle in women, taking medication, smoking and anti-COVID-19 vaccination
Experimentally validate the intrinsic performance | day 1
  Combined sensitivity and specificity measurements for all dogs according to canine characteristics (breed, age, experience) and canine detection procedures (start or end of line, test days, sequence effects).
Canine olfactory detection on mask | day 1
  High concordance kappa coefficient of detection performance between the respiratory mask and the sweat samples (axillary and/or neck).
Evaluation of the intrinsic and discriminative diagnostic performance of dogs for the olfactory detection of COVID-19 on sweat samples and/or used respiratory masks | day 1
  mesure combinée pour les chiens, d'une Sensibilité > 80%, d'une spécificité > 60% et des valeur prédictives positive et négative qui dépendront de la prévalence de la COVID-19 au sein de l'échantillon qui sera recruté consécutivement sans discrimination de sous-population

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PISTONE, Dr, Principal Investigator — University Hospital Bordeaux, France
Locations (6):
- France (6):
  - University Hospital Bordeaux, France, Bordeaux
  - Hospital Dax, Dax
  - Hospital Libourne, Libourne
  - University Hospital Limoges, France, Limoges
  - Hospital Périgueux, Périgueux
  - Universtity Hospital Poitiers, Poitiers